CLINICAL TRIAL: NCT01941706
Title: Preventing Depression in People With Epilepsy: an Extension of Project UPLIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: University of Michigan (Other); University of Washington (Other); The University of Texas Health Science Center, Houston (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Nancy J Thompson, PhD, Associate Professor, Behavioral Sciences and Health Education, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB00026786; 5RC1MD004563-02 (NIH); 09042433 (Other: Other)
Record Dates: First submitted 2013-09-05; First posted 2013-09-13 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Epilepsy; Depressive Symptoms; Depression; Seizure Disorder
Keywords: Epilepsy; Seizure; Cognitive Behavioral Therapy; Mindfulness; Depression; Depressive symptoms; prevention; Coping skills; Quality of life; Telehealth; Phone intervention; Internet-based intervention
MeSH Terms: conditions — Epilepsy; Depression; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Project UPLIFT (Treatment) (Experimental): Participants randomly assigned to the Treatment group receive the UPLIFT Intervention immediately after completing the Baseline Assessment. Participants can chose to participate in the Web- or phone-delivery of UPLIFT.
  Interventions: Behavioral: Project UPLIFT
- Project UPLIFT (TAU Waitlist Control) (Experimental): Participants randomly assigned to the Treatment-as Usual (TAU) Waitlist Control group will also receive the UPLIFT intervention. However, TAU Waitlist Control participants will begin the Intervention 8 weeks after completing the Baseline Assessment. During the initial 8 weeks, participants in this group will continue whatever treatment they are currently undergoing to prevent or treat mild depressive symptoms. Participants can chose to participate in the Web- or phone-delivery of UPLIFT.
  Interventions: Behavioral: Project UPLIFT

INTERVENTIONS:
Behavioral: Project UPLIFT — Developed for home-based treatment of depression in people with epilepsy, Project UPLIFT is based upon Mindfulness-based Cognitive Therapy for depression. It includes 8 modules, group-delivered by either telephone or Web. Trainees and people with epilepsy co-facilitate the groups, supervised by a licensed mental health professional.The co-facilitators are trained and supervised by the Principal Investigator, a Georgia-licensed clinical psychologist and Associate Professor of Behavioral Science and of Epidemiology in public health. Activities are designed to increase knowledge about depression; monitoring, challenging, and changing thoughts; coping and relaxing; attention and mindfulness; focusing on pleasure; the importance of reinforcement, and preventing relapse.

SUMMARY:
Project UPLIFT, a home-based treatment for depression in people with epilepsy, was designed to be delivered to groups by telephone or Web. The Project UPLIFT intervention materials were demonstrated to be effective in treating depression among people with epilepsy in Georgia. This project will assess whether the materials are also effective for preventing depression among people with epilepsy, and will extend the project beyond Georgia to Michigan, Texas, and Washington.

DETAILED DESCRIPTION:
The study is a pilot test of Project UPLIFT for depression prevention during which the acceptability and estimates of effectiveness of the intervention, presented in the Web and telephone modes, are assessed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of epilepsy
* at least three months post initial diagnosis of epilepsy and either on medication or permission of the physician
* symptoms of depression, but absence of moderate-to-severe depression, (8 < CES-D < 27)
* 21 years of age and older
* English speaking
* had access to a telephone
* mentally stable, as determined by a score of > 26 on the Telephone Mini-Mental Status Exam (T-MMSE)
* willing to participate
* willing to complete assessments three times

Exclusion Criteria:

* no diagnosis of epilepsy
* less than 3 months since diagnosis of epilepsy
* no depressive symptom (CES-D <8)
* severe depression (CES-D > 27)
* suicidal ideation
* previous participation in Project UPLIFT

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Changes in Depressive Symptoms | Baseline (at 0 week) , Interim (at 8 weeks), Follow-up (at16 weeks)
  Changes in depressive symptoms are measured using the modified Beck Depression Inventory (mBDI).

SECONDARY OUTCOMES:
Changes in seizure severity | Baseline (0 week), Interim (at 8 weeks), Follow-up (at 16 weeks)
  Changes in seizure severity measured using the Liverpool Seizure Severity.
Changes in Depression and Mindfulness Knowledge and Skills | Baseline (at 0 week), Interim (at 8 weeks), Follow-up (at 16 weeks)
  The changes are measured using an internally consistent scale assessing knowledge and skills associated with depression and mindfulness. The scale includes 18 true-false items assessing knowledge of depression based on the content of the UPLIFT modules. The scale also includes 13 Likert-scale assessing mindfulness skills based on the content of the UPLIFT modules.
Changes in Depressive Symptoms | baseline (at 0 week), Interim (at 8 weeks), Follow-up (at 16 weeks)
  Changes in depressive symptoms are measured using the Beck Depression Inventory (BDI).
Changes in Depressive Symptoms | baseline (at 0 week), Interim (at 8 weeks), Follow-up (at 16 weeks)
  Changes in depressive symptoms are measured using the Patient Health Questionnaire (PHQ-9).
Changes in Depressive Symptoms | baseline (at 0 week), Interim (at 8 weeks), Follow-up (at 16 weeks)
  Changes in depressive symptoms are measured using the Neurological Disorders Depression Inventory for Epilepsy (NDDI-E).
Change in Seizure Activity | Baseline (0 week), Interim (at 8 weeks), Follow-up (at 16 weeks)
  Change measured using self-reported number of seizures in the past 4 weeks.

OTHER OUTCOMES:
Changes in Satisfaction with Life | Baseline (at 0 week), Interim (at 8 weeks), Follow-up (at 16 weeks)
  Changes are measured using the Satisfaction with Life Scale (Denier, E., et al., The satisfaction with life scale. Journal of Personality Assessment, 1985)
Changes in Sleep Quality | Baseline (at 0 week), Interim (at 8 weeks), Follow-up (at 16 weeks)
  The study uses the Pittsburgh Sleep Quality Index to assess changes in sleep quality.
Changes in Depression Coping Self-Efficacy | Baseline (at 0 week), Interim (at 8 weeks), Follow-up (at 16 weeks)
  The study uses Perraud, S., Development of the Depression Coping Self-Efficacy Scale (DCSES). Archives of Psychiatric Nursing, 2000 to assess changes in depression coping self-efficacy.
Changes in Self Compassion | Baseline (at 0 week), Interim (at 8 weeks), Follow-up (at 16 weeks)
  The study uses Neff, K.D. and R. Vonk, Self-compassion versus global self-esteem: two different ways of relating to oneself. J Pers, 2009. 77(1): p. 23-50.. to assess changes in self compassion.
Changes in Physical and Mental Health Quality of Life | Baseline (at 0 week), Interim (at 8 weeks), Follow-up (at 16 weeks)
  The study uses the Centers for Disease Control's Behavioral Risk Factors Surveillance System (BRFSS) questionnaire to assess changes in physical and mental health quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Thompson, MPH, PhD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Rollins School of Public Health, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - University of Texas Health Science Center, Houston, Texas
  - University of Washington, Seattle, Washington